CLINICAL TRIAL: NCT03731377
Title: The Effectiveness of Mini-fluid Challenge in Predicting Fluid Responsiveness During Video Assisted Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 201807009RINC
Record Dates: First submitted 2018-10-01; First posted 2018-11-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Mini-fluid Challenge in Video-Assisted Thoracic Surgery
MeSH Terms: interventions — Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intubated group (Experimental): Patient in this group will receive general anesthesia with endotracheal tube intubation to perform one lung ventilation. Patient will be paralyzed and controlled ventilation will be implied.
  Interventions: Drug: Crystalloid Solutions
- Non-intubated group (Experimental): Patient in this group will receive general anesthesia with laryngeal mask insertion. Patients in this group will not be paralyzed and keep spontaneous breathing to maintain one lung ventilation.
  Interventions: Drug: Crystalloid Solutions

INTERVENTIONS:
Drug: Crystalloid Solutions — Mini-fluid challenge with crystalloid 250 ml will be given to patients first. After observation of hemodynamic parameters, further fluid challenge will be given for response observation.

SUMMARY:
Perioperative fluid management is crucial for patients' outcome. Muller et al developed a "Mini-fluid challenge method " to predict fluid responsiveness and the efficacy. The investigators design the study to investigate the effectiveness of mini-fluid challenge test in video assisted thoracic surgery.

DETAILED DESCRIPTION:
Perioperative fluid management is crucial for patients' outcome. Series of studies have indicated that adequate fluid management optimizes the cardiac out put, improves tissue perfusion, thus decrease the risk of postoperative morbidity. Muller et al developed a "Mini-fluid challenge method " to predict fluid responsiveness and the efficacy. Fluid status and proper perfusion condition in patients undergo thoracic surgery are especially crucial for the vulnerability of lung toward fluid overload. To the best of our knowledge, the efficacy of the test was not discussed in the perioperative care in video assisted thoracic surgery. The investigators design the study to investigate the effectiveness of mini-fluid challenge test in video assisted thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving scheduled video assisted thoracic surgery
* BMI 18.5~30 kg.m-2

Exclusion Criteria:

* age younger then 20 yrs or elder than 80 yrs
* pregnant women
* patients in intensive care units
* patients with the underlying disease including respiratory failure(FEV1/FVC < 70 % and FEV1 < 50%), heart failure(NYHA score =III、IV), kidney failure(eGFR< 60 ml.min-1.1.73m-2), liver failure
* patients with ongoing infection
* patient allergic to voluven

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-07 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure after fluid loading | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge

SECONDARY OUTCOMES:
Change of cardiac index after fluid loading | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge

OTHER OUTCOMES:
stroke volume variation(SVV) | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge
stroke volume (SV) | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge
stroke volume index(SVI) | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge
plethysmographic variation index(PVI) | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge
pulse pressure variation(PPV) | 3 hours
  Interpretate the correlation of mini-fluid challenge and conventional fluid challenge

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evans RG, Naidu B. Does a conservative fluid management strategy in the perioperative management of lung resection patients reduce the risk of acute lung injury? Interact Cardiovasc Thorac Surg. 2012 Sep;15(3):498-504. doi: 10.1093/icvts/ivs175. Epub 2012 May 22. PMID 22617510
- [Background] Cavallaro F, Sandroni C, Antonelli M. Functional hemodynamic monitoring and dynamic indices of fluid responsiveness. Minerva Anestesiol. 2008 Apr;74(4):123-35. Epub 2008 Jan 24. PMID 18212731
- [Background] Vincent JL. "Let's give some fluid and see what happens" versus the "mini-fluid challenge". Anesthesiology. 2011 Sep;115(3):455-6. doi: 10.1097/ALN.0b013e318229a521. No abstract available. PMID 21792055
- [Background] Wyffels PA, Sergeant P, Wouters PF. The value of pulse pressure and stroke volume variation as predictors of fluid responsiveness during open chest surgery. Anaesthesia. 2010 Jul;65(7):704-9. doi: 10.1111/j.1365-2044.2010.06371.x. Epub 2010 May 6. PMID 20477782